CLINICAL TRIAL: NCT04516759
Title: A Phase II, Randomised, Double-blind, Placebo-controlled Clinical Trial to Assess the Safety and Efficacy of AZD1656 in Diabetic Patients Hospitalised With Suspected or Confirmed COVID-19
Brief Title: AZD1656 in Diabetic Patients Hospitalised With Suspected or Confirmed COVID-19
Acronym: ARCADIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St George Street Capital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SGS.1656.201; 2020-002211-21 (EudraCT Number)
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Results first posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Covid19
Keywords: COVID-19; Diabetes Mellitus; SARS-CoV-2; Regulatory T Cell; Glucokinase
MeSH Terms: conditions — COVID-19; Diabetes Mellitus; Maturity-Onset Diabetes of the Young, Type 2 | interventions — AZD1656

STUDY DESIGN:
Intervention Model Description: This is a randomised double-blind study. Eligible patients will be randomly assigned to one of two groups (AZD1656 plus usual care or placebo plus usual care) on a 1:1 basis
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AZD1656 (plus Usual Hospital Care) (Experimental): 50mg film-coated tablets at a dose of 100mg BID
  Interventions: Drug: AZD1656
- Matched Placebo (plus Usual Hospital Care) (Placebo Comparator): Matched placebo tablets
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AZD1656 — 50mg film-coated tablets (at daily dose of 100mg BID)
  Arms: AZD1656 (plus Usual Hospital Care)
Other: Placebo — Matched placebo tablets
  Arms: Matched Placebo (plus Usual Hospital Care)

SUMMARY:
The ARCADIA Trial is a randomised, double-blind, placebo-controlled clinical trial to assess the safety and efficacy of AZD1656 in patients with either Type 1 or Type 2 diabetes, hospitalised with COVID-19.

DETAILED DESCRIPTION:
The ARCADIA Trial will assess the safety and efficacy of AZD1656 in 150 patients with either Type 1 or Type 2 diabetes who have been hospitalised with COVID-19.

AZD1656 is a glucokinase (GK; hexokinase 4) activator which has been shown to reduce blood glucose for up to 4 months in humans. Diabetic patients admitted to hospital with COVID-19 often present with hyperglycaemia and are particularly vulnerable to progression to severe COVID-19. Treatment with AZD1656 (in addition to their usual care) may provide additional glucose control which could help improve clinical outcomes in both Type 1 and Type 2 diabetic populations.

In addition to its glucose lowering effect, AZD1656 may have additional benefits to COVID-19 patients via its effects on immune function. In many patients with severe COVID-19, an overreaction of the body's own immune system can cause severe problems including damage to the lungs and heart, which can lead to breathing problems necessitating intubation and ventilation. AZD1656 has been shown to activate the migration of T regulatory cells to sites of inflammation in preclinical experiments. This migration of Treg cells to inflamed tissue is crucial for their immune-modulatory function (Kishore et al (2017)). AZD1656 could enhance Treg migratory capacity and may prevent the development of cardiorespiratory complications observed in hospitalised patients with COVID-19, leading to lower requirements for oxygen therapy and assisted ventilation, and reduced incidences of pneumonia and acute respiratory distress syndrome (ARDS).

Diabetic patients hospitalised with COVID-19 will be randomised to receive either AZD1656 tablets or placebo tablets on a 1:1 basis until they are discharged from hospital or until they require intubation/mechanical ventilation. The aim of the study is to determine whether AZD1656 improves clinical outcomes in diabetic patients hospitalised with COVID-19. The World Health Organization (WHO) 8-point Ordinal Scale for Clinical Improvement will be used as the standard methodology for measuring patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female.
2. Aged 18 and older.
3. Have either Type I or Type II Diabetes Mellitus.
4. Hospitalised with suspected or confirmed novel coronavirus (Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)) infection at time of enrolment, categorised as stage 3, 4 or 5 on the WHO Ordinal Scale for Clinical Improvement.
5. Blood glucose level at or above 4 mmol/L.
6. Able to take oral (tablet) formulation of medication.
7. Patient is able to provide written informed consent prior to initiation of any study procedures.

Exclusion Criteria:

1. In the opinion of the clinical team, progression to intubation or mechanical ventilation is imminent and inevitable, within the next 24 hours, irrespective of the provision of treatments.
2. Patients admitted with primary suspected or proven Mycoplasma pneumoniae, Chlamydia pneumoniae and bacterial pneumonia, who acquired COVID-19 while hospitalized.
3. Treatment with immunomodulators or anti-rejection drugs within the last 3 months.
4. Pregnant or breast feeding.
5. Men, and women of child-bearing potential, unwilling to use highly effective contraception during their participation in the trial and for 2 weeks after study completion.
6. Anticipated transfer to another hospital which is not a study site within 72 hours.
7. Known sensitivity to any of the study medication/placebo excipients.
8. Prior dosing with AZD1656 on a previous clinical trial.
9. Patients admitted as a result of and receiving immediate treatment for an acute asthmatic attack, acute myocardial infarction, acute cerebrovascular event.
10. Any known non-COVID-19, non-diabetes related, serious condition which, in the opinion of the clinical team, makes the patient unsuitable for the trial.
11. Known history of drug or alcohol abuse within previous 12 months of screening.
12. Known history of HIV, hepatitis C or unresolved hepatitis B or severe liver disease.
13. Current or planned use of gemfibrozil or any other strong inhibitors of CYP2C8.
14. Current or previous participation in another clinical trial where the patient has received a dose of an Investigational Medicinal Product (IMP) containing small molecule treatment(s) within 30 days or 5 half-lives (whichever is longer) prior to enrolment into this study, or containing biological treatment(s) within 3 months prior to entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-04-25 (Actual); Study Completion 2021-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kieran McCafferty, MD, Principal Investigator — Barts & The London NHS Trust
Locations (30):
- Czechia (7):
  - Masarykova Univerzita - Fakultni Nemocnice U SV Anny V Brne (308), Brno
  - Nemocnice Hořovice (309), Hořovice
  - Oblastni Nemocnice Kolín (306), Kolín
  - Klaudianova Nemonice (302), Mladá Boleslav
  - Fakultni Nemocnice V Motole (303), Prague
  - Thomayerova Nemonice (310), Prague
  - Nemocnice Třebíč (305), Třebíč
- Romania (8):
  - Colentina Clinical Hospital (204), Bucharest
  - Spitalul Clinic de Boli Infectioase Cluj-Napoca (203), Cluj-Napoca
  - Spitalul Clinic de Pneumoftiziologie "Leon Daniello" Cluj-Napoca (202), Cluj-Napoca
  - Spitalul Clinic de Boli Infectioase Constanţa (207), Constanța
  - Spitalul Clinic de Boli Infectioase si Pneumoftiziologie Dr Victor Babes Craiova (206), Craiova
  - Spitalul Judetean de Urgenta Deva (208), Deva
  - Spitalul Clinic de Boli Infectioase "Sfanta Parascheva" Iaşi (205), Iași
  - Spitalul Clinic de Boli Infectioase si Pneumoftiziologie Dr Victor Babes Timişoara (201), Timișoara
- United Kingdom (15):
  - Barnsley Hospital NHS Foundation Trust (105), Barnsley
  - Bolton NHS Foundation Trust (122), Bolton
  - Bradford Teaching Hospitals NHS Foundation Trust (103), Bradford
  - North Bristol NHS Trust (116), Bristol
  - County Durham and Darlington NHS Foundation Trust (121), Darlington
  - The Dudley Group NHS Foundation Trust (107), Dudley
  - Medway NHS Foundation Trust (108), Gillingham
  - Hull & East Yorkshire NHS Trust (102), Hull
  - Barts Health NHS Trust (101 and 111), London
  - Royal Free London NHS Foundation Trust (119), London
  - St George's University Hospitals NHS Foundation Trust (114), London
  - Penine Acute Hospitals NHS Trust (106), Salford
  - Sheffield Hospitals NHS Foundation Trust (104), Sheffield
  - Somerset NHS Foundation Trust (109), Taunton
  - Walsall Healthcare NHS Trust (113), Walsall

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to deidentified individual participant data (IDP) that underlie the published clinical trial results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Requests for access to the data will be accepted beginning 6 months after article publication and will continue to be accepted for up to 5 years after publication.
Access Criteria: Researchers must submit a methodologically sound research proposal to St George Street using the contact details provided on our website. See link below.
URL: http://www.sgscapital.org

REFERENCES:
- [Derived] Chorlton J, Hollowood Z, Dyer C, Lockhart D, Boekman P, McCafferty K, Coffey P, Marelli-Berg F, Martin J. A randomised, double-blind, placebo-controlled, multicentre clinical trial of AZD1656 in diabetic patients hospitalised with COVID-19: The ARCADIA Trial - implications for therapeutic immune modulation. EClinicalMedicine. 2022 Sep;51:101604. doi: 10.1016/j.eclinm.2022.101604. Epub 2022 Aug 18. PMID 35996565
- [Derived] McCafferty K, Hollowood Z, Allen M, Lockhart D, Chorlton J, Martin J. ARCADIA study protocol: a phase II, randomised, double-blind, placebo-controlled clinical trial to assess the safety and efficacy of AZD1656 in patients with diabetes hospitalised with suspected or confirmed COVID-19. BMJ Open. 2021 Dec 1;11(12):e049650. doi: 10.1136/bmjopen-2021-049650. PMID 34853102

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 170 subjects were screened for participation. 13 subjects were screening failures. 156 subjects were randomized of which 3 subjects withdrew consent prior to start of study medication. 153 subjects started with study treatment.
Period: Overall Study
Arm/Group | AZD1656 (Plus Usual Hospital Care) | Matched Placebo (Plus Usual Hospital Care)
Started | 80 (excluding 2 subjects who were randomized but did not start treatment) | 73 (excluding 1 subject who was randomized but did not start treatment)
Completed | 79 | 71
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD1656 (Plus Usual Hospital Care) | Matched Placebo (Plus Usual Hospital Care) | Total
Number analyzed (Participants) | 80 | 73 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 31 | 69
  >=65 years | 42 | 42 | 84
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 26 | 56
  Male | 50 | 47 | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 77 | 70 | 147
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 19 | 14 | 33
  Czechia | 27 | 22 | 49
  United Kingdom | 34 | 37 | 71
WHO OSCI rating [Count of Participants; unit: Participants] — Patients hospitalised with suspected or confirmed novel coronavirus (SARSCoV-2) infection, categorised as 3, 4 or 5 on the WHO Ordinal Scale for Clinical Improvement, were considered eligible for the trial. This score was clinically assessed by the treating physician at baseline. The WHO score ranges from 0-8 (0 = no symptoms, 8 = death). The higher the score the worse the condition of the patient is/was.
  Participants
    3 - Hospitalised, no oxygen | 19 | 13 | 32
    4 - Hospitalised, oxygen | 52 | 42 | 94
    5 - Non-invasive ventilation or high flow oxygen | 9 | 18 | 27
Diabetes Type [Count of Participants; unit: Participants]
  Type 1 | 1 | 2 | 3
  Type 2 | 79 | 71 | 150
Vitamin D group [Count of Participants; unit: Participants]
  < 25 nmol/l | 31 | 27 | 58
  >= 25 nmol/l | 46 | 45 | 91
  missing | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Clinical Improvement by Day 14
Description: The World Health Organization (WHO) 8-point Ordinal Scale for Clinical Improvement (OSCI) was used to measure Clinical Improvement at Day 14 versus baseline, comparing AZD1656 treatment with placebo. The WHO OSCI score ranges from 0-8 (0 = no symptoms, 8 = death). The higher the score the worse the condition of the patient.
  Results are presented as number of responders. Patients who were assigned a WHO score of 1, 2 or 3 at Day 14 were considered a treatment responder. A patient who was discharged before Day 14 was also considered a responder. All other patients (WHO scores 4-8 at Day 14) were considered treatment failures.
Time Frame: Day 1 to Day 14
Population: Full Analysis Set: all participants who received at least one dose of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | AZD1656 (Plus Usual Hospital Care) | Matched Placebo (Plus Usual Hospital Care)
Number analyzed (Participants) | 80 | 73
Participants
  Treatment responder | 61 | 51
  Treatment failure | 18 | 21
  Missing | 1 | 1
Statistical Analysis 1: Comparison: AZD1656 (Plus Usual Hospital Care) vs Matched Placebo (Plus Usual Hospital Care); Test type: Superiority; p = 0.1854, Chi-squared; Chi-squared test on the one-sided significance level of 2.5%; Risk Ratio (RR) = 1.09, 95% CI 2-sided [0.9 to 1.32]

2. Secondary Outcome: Clinical Improvement at Day 7, 14 and 21
Description: The World Health Organization (WHO) 8-point Ordinal Scale for Clinical Improvement (OSCI) was used to measure Clinical Improvement at Day 7, Day 14 and Day 21 versus baseline, comparing AZD1656 treatment with placebo.
  Results are presented as the percentage of patients categorised at each severity rating at each timepoint on the WHO 8-point OSCI scale.
  The WHO OSCI score ranges from 0-8 (0 = no symptoms, 8 = death). The higher the score the worse the condition of the patient.
  Study Drug Discontinuation was the date on which a patient discontinued treatment. Treatment was given for a maximum of 21 days, or until date of hospital discharge (WHO score 1 or 2), or date mechanical ventilation was required (WHO score 6 or 7) or until date of death (WHO score 8).
Time Frame: Day 1 to Day 21
Population: Full Analysis Set: all participants who received at least one dose of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | AZD1656 (Plus Usual Hospital Care) | Matched Placebo (Plus Usual Hospital Care)
Number analyzed (Participants) | 80 | 73
Participants
  Baseline: Score 1: Ambulatory - no limitation of activities | 0 | 0
  Baseline: Score 2: Ambulatory - limitation of activities | 0 | 0
  Baseline: Score 3: Hospitalized, no oxygen therapy | 19 | 13
  Baseline: Score 4: Hospitalized, oxygen by mask or nasal prongs | 52 | 42
  Baseline: Score 5: Hospitalized, non-invasive ventilation or high-flow oxygen | 9 | 18
  Baseline: Score 6: Hospitalized, intubation or mechanical ventilation | 0 | 0
  Baseline: Score 7: Hospitalized, ventilation + additional organ support - pressors, RTT, ECMO | 0 | 0
  Baseline: Score 8: Death | 0 | 0
  Baseline: Missing | 0 | 0
  Day 7: Score 1: Ambulatory - no limitation of activities | 7 | 7
  Day 7: Score 2: Ambulatory - limitation of activities | 22 | 10
  Day 7: Score 3: Hospitalized, no oxygen therapy | 15 | 17
  Day 7: Score 4: Hospitalized, oxygen by mask or nasal prongs | 23 | 26
  Day 7: Score 5: Hospitalized, non-invasive ventilation or high-flow oxygen | 10 | 5
  Day 7: Score 6: Hospitalized, intubation or mechanical ventilation | 2 | 3
  Day 7: Score 7: Hospitalized, ventilation + additional organ support - pressors, RTT, ECMO | 0 | 0
  Day 7: Score 8: Death | 0 | 5
  Day 7: Missing | 1 | 0
  Day 14: Score 1: Ambulatory - no limitation of activities | 16 | 14
  Day 14: Score 2: Ambulatory - limitation of activities | 37 | 30
  Day 14: Score 3: Hospitalized, no oxygen therapy | 8 | 7
  Day 14: Score 4: Hospitalized, oxygen by mask or nasal prongs | 9 | 10
  Day 14: Score 5: Hospitalized, non-invasive ventilation or high-flow oxygen | 4 | 2
  Day 14: Score 6: Hospitalized, intubation or mechanical ventilation | 4 | 3
  Day 14: Score 7: Hospitalized, ventilation + additional organ support - pressors, RTT, ECMO | 0 | 0
  Day 14: Score 8: Death | 1 | 6
  Day 14: Missing | 1 | 1
  Day 21: Score 1: Ambulatory - no limitation of activities | 20 | 15
  Day 21: Score 2: Ambulatory - limitation of activities | 44 | 41
  Day 21: Score 3: Hospitalized, no oxygen therapy | 4 | 0
  Day 21: Score 4: Hospitalized, oxygen by mask or nasal prongs | 2 | 5
  Day 21: Score 5: Hospitalized, non-invasive ventilation or high-flow oxygen | 4 | 2
  Day 21: Score 6: Hospitalized, intubation or mechanical ventilation | 4 | 3
  Day 21: Score 7: Hospitalized, ventilation + additional organ support - pressors, RTT, ECMO | 0 | 0
  Day 21: Score 8: Death | 1 | 6
  Day 21: Missing | 1 | 1
  Study Drug Discontinuation (SDD): Score 1: Ambulatory - no limitation of activities | 20 | 15
  Study Drug Discontinuation (SDD): Score 2: Ambulatory - limitation of activities | 44 | 40
  Study Drug Discontinuation (SDD): Score 3: Hospitalized, no oxygen therapy | 3 | 0
  Study Drug Discontinuation (SDD): Score 4: Hospitalized, oxygen by mask or nasal prongs | 3 | 5
  Study Drug Discontinuation (SDD): Score 5: Hospitalized, non-invasive ventilation or high-flow oxygen | 4 | 1
  Study Drug Discontinuation (SDD): Score 6: Hospitalized, intubation or mechanical ventilation | 4 | 3
  Study Drug Discontinuation (SDD): Score 7: Hospitalized, ventilation + additional organ support - pressors, RTT, ECMO | 0 | 0
  Study Drug Discontinuation (SDD): Score 8: Death | 1 | 6
  Study Drug Discontinuation (SDD): Missing | 1 | 3
Statistical Analysis 1: Comparison: AZD1656 (Plus Usual Hospital Care) vs Matched Placebo (Plus Usual Hospital Care); Test type: Other; p = 0.0286, Wilcoxon (Mann-Whitney) — Baseline p-value; one-side significance level of 2.5%
Statistical Analysis 2: Comparison: AZD1656 (Plus Usual Hospital Care) vs Matched Placebo (Plus Usual Hospital Care); Test type: Other; p = 0.0786, Wilcoxon (Mann-Whitney) — Day 7 p-value; one-side significance level of 2.5%
Statistical Analysis 3: Comparison: AZD1656 (Plus Usual Hospital Care) vs Matched Placebo (Plus Usual Hospital Care); Test type: Other; p = 0.2169, Wilcoxon (Mann-Whitney) — Day 14 p-value; one-side significance level of 2.5%
Statistical Analysis 4: Comparison: AZD1656 (Plus Usual Hospital Care) vs Matched Placebo (Plus Usual Hospital Care); Test type: Other; p = 0.1860, Wilcoxon (Mann-Whitney) — Day 21 p-value; one-sided significance level of 2.5%
Statistical Analysis 5: Comparison: AZD1656 (Plus Usual Hospital Care) vs Matched Placebo (Plus Usual Hospital Care); Test type: Other; p = 0.2256, Wilcoxon (Mann-Whitney) — Study Drug Discontinuation (SDD) p-value; one-sided significance level of 2.5%

3. Secondary Outcome: Glycaemic Control
Description: Degree of glycaemic control as measured by the need to increase baseline medication requirements or the need to add additional diabetic medications to maintain appropriate blood glucose levels in patients receiving AZD1656 compared with placebo
Time Frame: Day 1 to Day 21
Population: Full Analysis Set: all participants who at least received one dose of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | AZD1656 (Plus Usual Hospital Care) | Matched Placebo (Plus Usual Hospital Care)
Number analyzed (Participants) | 80 | 73
Participants
  Increase in Diabetic Medication Needed equal or More Than 3 Days: True | 12 | 13
  Increase in Diabetic Medication Needed equal or More Than 3 Days: False | 68 | 60
  Diabetic Medication is Stable/Reduced Equal or More Than 3 days: True | 61 | 58
  Diabetic Medication is Stable/Reduced Equal or More Than 3 days: False | 19 | 15
  Increase in Diabetic Medication Needed at Any Time During the Study: True | 25 | 21
  Increase in Diabetic Medication Needed at Any Time During the Study: False | 55 | 52
  Diabetic Medication is Stable/Reduced at Any Time During the Study: True | 74 | 67
  Diabetic Medication is Stable/Reduced at Any Time During the Study: False | 6 | 6
Statistical Analysis 1: Comparison: AZD1656 (Plus Usual Hospital Care) vs Matched Placebo (Plus Usual Hospital Care); Test type: Other; p = 0.4006, Fisher Exact — Increase in Diabetic Medication needed equal or more than 3 days
Statistical Analysis 2: Comparison: AZD1656 (Plus Usual Hospital Care) vs Matched Placebo (Plus Usual Hospital Care); Test type: Other; p = 0.7482, Fisher Exact — Diabetic Medication is stable/reduced equal or more than 3 days
Statistical Analysis 3: Comparison: AZD1656 (Plus Usual Hospital Care) vs Matched Placebo (Plus Usual Hospital Care); Test type: Other; p = 0.6949, Fisher Exact — Increase in Diabetic Medication needed at any time during the study
Statistical Analysis 4: Comparison: AZD1656 (Plus Usual Hospital Care) vs Matched Placebo (Plus Usual Hospital Care); Test type: Other; p = 0.5521, Fisher Exact — Diabetic Medication is stable/reduced at any time during the study

4. Secondary Outcome: Occurrence of Adverse Events
Description: Proportion of Treatment Emergent Adverse Events (TEAEs) leading to study drug discontinuation in patients receiving AZD1656 compared with placebo
Time Frame: Day 1 to Day 28
Population: This analysis includes all participants who received at least one dose of treatment and had at least one post-baseline safety assessment (where the statement that a patient had no AE on the AE eCRF constitutes a safety assessment). 4 patients from the placebo arm are moved to the AZD1656 arm due to having drug in their PK samples. The assignment of patients to the treatment groups are as actually treated.
Measure: Number; unit: Events
Arm/Group | AZD1656 (Plus Usual Hospital Care) | Matched Placebo (Plus Usual Hospital Care)
Number analyzed (Participants) | 84 | 69
Events
  TEAEs leading to study drug discontinuation | 2 | 2
  Other TEAEs | 28 | 21
Statistical Analysis 1: Comparison: AZD1656 (Plus Usual Hospital Care) vs Matched Placebo (Plus Usual Hospital Care); Test type: Other; p = 0.5875, Fisher Exact

5. Secondary Outcome: Occurrence of Serious Adverse Events
Description: Proportion of Serious Adverse Events (SAEs) in patients receiving AZD1656 compared with placebo
Time Frame: Day 1 to Day 28
Population: This analysis includes all patients who received at least one dose of IMP and had at least one post-baseline safety assessment (where the statement that a patient had no AE on the AE eCRF constitutes a safety assessment). 4 patients from the placebo arm are moved to the AZD1656 arm due to having drug in their PK samples. The assignment of patients to the treatment groups are as actually treated.
Measure: Number; unit: Events
Arm/Group | AZD1656 (Plus Usual Hospital Care) | Matched Placebo (Plus Usual Hospital Care)
Number analyzed (Participants) | 84 | 69
Events
  Serious Adverse Events | 4 | 7
  Other AEs | 28 | 17
Statistical Analysis 1: Comparison: AZD1656 (Plus Usual Hospital Care) vs Matched Placebo (Plus Usual Hospital Care); Test type: Other; p = 0.1129, Fisher Exact

6. Secondary Outcome: Duration of Hospitalisation
Description: Time from hospital admission to hospital discharge (in hours) in patients receiving AZD1656 compared with placebo
Time Frame: Day 1 to Day 21
Population: Full Analysis Set: all participant who at least received on dose of treatment
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | AZD1656 (Plus Usual Hospital Care) | Matched Placebo (Plus Usual Hospital Care)
Number analyzed (Participants) | 80 | 73
hours | 264.3 [215.5 to 299.7] | 288.7 [260.1 to 307.1]
Statistical Analysis 1: Comparison: AZD1656 (Plus Usual Hospital Care) vs Matched Placebo (Plus Usual Hospital Care); Test type: Superiority; p = 0.1556, Log Rank

7. Secondary Outcome: Mortality Rate
Description: Mortality rate in patients receiving AZD1656 compared with placebo.
Time Frame: Day 1 to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | AZD1656 (Plus Usual Hospital Care) | Matched Placebo (Plus Usual Hospital Care)
Number analyzed (Participants) | 80 | 73
Participants
  Died | 4 | 9
  Did not die | 75 | 63
  Missing | 1 | 1
Statistical Analysis 1: Comparison: AZD1656 (Plus Usual Hospital Care) vs Matched Placebo (Plus Usual Hospital Care); Test type: Other; p = 0.0903, Fisher Exact; The p-value is assessed by means of an Fisher's exact test on the one-sided significance level of 2.5%; Risk Ratio (RR) = 0.41, 95% CI 2-sided [0.13 to 1.26]

8. Secondary Outcome: Intubation/Mechanical Ventilation
Description: Number of Patients Receiving Intubation/Mechanical Ventilation
Time Frame: Day 1 to Day 21
Population: Full Analysis Set: all participants who at least received one dose of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | AZD1656 (Plus Usual Hospital Care) | Matched Placebo (Plus Usual Hospital Care)
Number analyzed (Participants) | 80 | 73
Participants
  Receiving Intubation/Mechanical Ventilation | 3 | 3
  Not Receiving Intubation/Mechanical Ventilation | 76 | 69
  Missing | 1 | 1
Statistical Analysis 1: Comparison: AZD1656 (Plus Usual Hospital Care) vs Matched Placebo (Plus Usual Hospital Care); Test type: Other; p = 0.6144, Fisher Exact; One-sided significance level of 2.5%

9. Post Hoc Outcome: Mortality Rate
Description: Mortality rate from randomization up to and including 168 hours post randomization
Time Frame: Randomization to 168 hours post randomization
Population: Full Analysis Set: all participant who received at least one dose of treatment; patients who withdrew consent are categorised as missing
Measure: Count of Participants; unit: Participants
Arm/Group | AZD1656 (Plus Usual Hospital Care) | Matched Placebo (Plus Usual Hospital Care)
Number analyzed (Participants) | 80 | 73
Participants
  Died | 0 | 6
  Did not die | 79 | 66
  Missing | 1 | 1
Statistical Analysis 1: Comparison: AZD1656 (Plus Usual Hospital Care) vs Matched Placebo (Plus Usual Hospital Care); Test type: Other; p = 0.0105, Fisher Exact; one-sided significance level of 2.5%

10. Post Hoc Outcome: Proportion of Patients Discharged up to and Including 168 Hours Having a WHO OSCI Rating of 1 or 2
Description: Proportion of Patients Being Discharged From Hospital up to and Including 168 hrs Having WHO OSCI Rating of 1 or 2
Time Frame: Day 1 up to and including 168 hours post randomization
Population: Full Analysis Set: all participants who had at least one dose of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | AZD1656 (Plus Usual Hospital Care) | Matched Placebo (Plus Usual Hospital Care)
Number analyzed (Participants) | 80 | 73
Participants
  Discharged from hospital (within 168 hrs with WHO 1 or 2) | 30 | 18
  Not discharged from Hospital (within 168 hrs with WHO 1 or 2) | 49 | 54
  Missing | 1 | 1
Statistical Analysis 1: Comparison: AZD1656 (Plus Usual Hospital Care) vs Matched Placebo (Plus Usual Hospital Care); Test type: Other; p = 0.062, Fisher Exact; one-sided significance level of 2.5%

ADVERSE EVENTS:
Time Frame: All AEs, including SAEs, were captured after signing the informed consent and until 7 days after treatment discontinuation (up to a maximum of 28 days).
Description: Serious and other Adverse Events were assessed using the Safety Set (SAF) dataset. The SAF dataset included 84 patients in the AZD1656 arm and 69 patients in the placebo arm, All-Cause Mortality was assessed using the Full Analysis Set (FAS) dataset. The FAS dataset included 80 patients in the AZD1656 arm and 73 patients in the placebo arm.
Arm/Group | AZD1656 (Plus Usual Hospital Care) | Matched Placebo (Plus Usual Hospital Care)
All-Cause Mortality (participants affected / at risk) | 4/80 | 9/73
Serious Adverse Events (participants affected / at risk) | 10/84 | 19/69
Other Adverse Events (participants affected / at risk) | 43/84 | 17/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD1656 (Plus Usual Hospital Care) (N=84) | Matched Placebo (Plus Usual Hospital Care) (N=69)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Abcess limb (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 5 (5)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) — Sepsis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD1656 (Plus Usual Hospital Care) (N=84) | Matched Placebo (Plus Usual Hospital Care) (N=69)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Vitamin D decreased (Investigations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Leucocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Reversible ischaemic neurological deficit (Nervous system disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 8 (13) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Oral fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT04516759/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT04516759/SAP_001.pdf